CLINICAL TRIAL: NCT03799822
Title: Safety and Efficacy of Vitamin K Antagonists Versus Rivaroxaban in Hemodialysis Patients With Atrial Fibrillation: a Multicenter Randomized Controlled Trial
Brief Title: Oral Anticoagulation in Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Rogier Caluwe, Principal Investigator, Onze Lieve Vrouw Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OLV 2014/065
Record Dates: First submitted 2019-01-07; First posted 2019-01-10 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Atrial Fibrillation
Keywords: hemodialysis; rivaroxaban; vitamin K2
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Active Comparator): Hemodialysis patients with non valvular atrial fibrillation receiving warfarin
  Interventions: Drug: Vitamin K Antagonist - Drug
- rivaroxaban (Experimental): Hemodialysis patients with non valvular atrial fibrillation receiving rivaroxaban 10 mg od
  Interventions: Drug: Rivaroxaban 10 MG Oral Tablet
- rivaroxaban + K2 (Experimental): Hemodialysis patients with non valvular atrial fibrillation receiving rivaroxaban 10 mg od + vitamin K2 supplements
  Interventions: Drug: Rivaroxaban 10 MG Oral Tablet; Dietary Supplement: MK-7 2000µg thrice weekly

INTERVENTIONS:
Drug: Rivaroxaban 10 MG Oral Tablet — replacement of warfarin by rivaroxaban
  Arms: rivaroxaban; rivaroxaban + K2
Dietary Supplement: MK-7 2000µg thrice weekly — dietary supplement of vitamin K2 MK-7 2000µg thrice weekly
  Arms: rivaroxaban + K2
Drug: Vitamin K Antagonist - Drug — treatment with a vitamin K antagonist
  Arms: Control

SUMMARY:
The investigators refer to the trial with clinicaltrials.gov indentifier NCT02610933 entitled Effect on Vascular Calcification of Replacing Warfarin by Rivaroxaban With or Without VitK2 in Hemodialysis Patients.

After termination of this trial, included patients will be asked to participate in the extension trial by continuing the treament of their respective allocation arm. No new intervention will be done.

DETAILED DESCRIPTION:
The investigators refer to the trial with clinicaltrials.gov indentifier NCT02610933 entitled Effect on Vascular Calcification of Replacing Warfarin by Rivaroxaban With or Without VitK2 in Hemodialysis Patients.

After termination of this trial, included patients will be asked to participate in the extension trial by continuing the treament of their respective allocation arm. No new intervention will be done. Relevant endpoints like death, cardiovascular events and bleeding episodes will be registered.

ELIGIBILITY:
Inclusion Criteria:

* inclusion in the trial with clinicaltrials.gov identifier NCT02610933
* signed informed consent for this extension trial

Exclusion Criteria:

* none

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
composite of fatal and non-fatal stroke and other cardiovascular events | through study completion, on average 3 years
  composite of fatal and non-fatal stroke and other cardiovascular events

SECONDARY OUTCOMES:
death rate | through study completion, on average 3 years
  cause of death
safety: incidence of life-threatening, major and minor bleeding | through study completion, on average 3 years
  incidence of life-threatening, major and minor bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Rogier Caluwe, MD, Principal Investigator — OLV Hospital Aalst, Belgium
Locations (1):
- OLV Hospital, Aalst, Belgium

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593
- [Derived] De Vriese AS, Caluwe R, Van Der Meersch H, De Boeck K, De Bacquer D. Safety and Efficacy of Vitamin K Antagonists versus Rivaroxaban in Hemodialysis Patients with Atrial Fibrillation: A Multicenter Randomized Controlled Trial. J Am Soc Nephrol. 2021 Jun 1;32(6):1474-1483. doi: 10.1681/ASN.2020111566. Epub 2021 Mar 22. PMID 33753537